CLINICAL TRIAL: NCT02511652
Title: Comparison of the Ambu AuraGain vs. LMA Supreme in Paralysed Patients Undergoing Gynecologic Laparoscopic Surgery in the Trendelemburg Position
Brief Title: Ambu AuraGain vs LMA Supreme in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Ana M Lopez, MD, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBarcelona
Record Dates: First submitted 2015-07-20; First posted 2015-07-30 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Laparoscopy; Airway Management; Supraglottic Airway Devices
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambu AuraGain (Active Comparator): Insertion of the supraglottic device and evaluation of its clinical performance
  Interventions: Device: Ambu AuraGain evaluation; Procedure: Laparoscopic surgery
- LMA Supreme (Active Comparator): Insertion of the supraglottic device and evaluation of its clinical performance
  Interventions: Device: LMA Supreme evaluation; Procedure: Laparoscopic surgery

INTERVENTIONS:
Device: Ambu AuraGain evaluation — Evaluation of clinical performance in terms of Insertion, ventilation, position and complications
  Arms: Ambu AuraGain
Device: LMA Supreme evaluation — Evaluation of clinical performance in terms of Insertion, ventilation, position and complications
  Arms: LMA Supreme
Procedure: Laparoscopic surgery — Gynecologic laparoscopic surgery in the trendelemburg position

SUMMARY:
The aim of the study is to compare the performance of two supraglottic airway devices (SGA), the new Ambu AuraGain and the LMA Supreme, in sixty female patients undergoing gynaecologic laparoscopy in the trendelemburg position.

Primary outcome is the airway seal pressure. Secondary outcomes are ease of insertion, quality of ventilation, endoscopic view of the glottis, gastric tube passage and complications.

DETAILED DESCRIPTION:
The patients are randomly assigned to 2 groups:

* Group 1: Ambu AuraGain.
* Group 2: LMA Supreme, Teleflex

Procedure:

The investigation protocol contains the following sections:

1. Induction of anaesthesia. Intravenous infusion of remifentanil and propofol targeting the effect site (2-4 ng/ml and 4-6 µg/ml respectively). No muscle relaxant will be used for insertion of the SGA. Rocuronium 0.2 mg/Kg will be administered before initiation of pneumoperitoneum.
2. Insertion of the SGAs. The size of the SGA device used is based on the manufacturers' recommendations. All devices are deflated a lubricated prior to use. Once inserted, the cuff is be inflated with a manometer up to 60 cm H20 Position of the device is adjusted if needed. Data recorded: size of SGA, time an number of attempts.
3. Fibreoptic evaluation of the SGAs anatomical position: complete view of the vocal cords (I), epiglottis visible inside, but not causing obstruction (II), epiglottis visible and obstructing the glottic inlet (III), or glottic structures not identified (IV).
4. Functionality of the gastric drainage channel of the SGAs: passage of a 16 G size tube.
5. Measurement of airway seal pressure (oropharyngeal leak pressure (OLP): at baseline, and at 15, 30 and 60 minutes. The maximum pressure allowed is 40 cm H2O.
6. Ventilatory mechanics and parameters are measured at baseline, and at 15, 30 and 60 minutes.

   Perioperative complications: Hiccup, gastric distension, regurgitation / Aspiration, airway obstruction, laryngospasm, dental, mucosal or tongue injury, hypoxia (SpO2 < 92%)
7. Removal of the SGAs: Presence of blood - 3 level grading (+/++/+++) Postoperative complications: sore throat, hoarseness, dysphonia, dysphagia, dysphagia: 3-point scale

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated as eligible for a SGA
* ASA I-III
* Without criteria for difficult airway
* Body Mass Index ≤ 35 kg/m2
* The patient has signed the Informed Consent
* The patient understands his or hers rights and consequences related to this investigation

Exclusion Criteria:

* Planned operation time > 2 hours
* High risk of regurgitation
* Respiratory tract pathology
* Preoperative sore throat
* Patients with a known or predicted difficult airway
* Patients diagnosed with dementia or any mental handicaps
* Patient who has a guardian.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Airway seal pressure | At 15 minutes
  Maximum airway pressure that the device can achieve without oropharyngeal leak of gas.

SECONDARY OUTCOMES:
Ease of insertion of the device | Baseline
  Time needed to insert the device
Change in Quality of ventilation | At baseline and at 15, 30 and 60 minutes
  number of manoeuvres/corrections required
Endoscopic view of glottic structures | At 15 minutes
  Assessment of alignment with the glottic inlet as: complete view of the vocal cords (I), epiglottis visible inside, but not causing any obstruction (II), epiglottis visible and causing obstruction (III) or glottis not identified (IV)
Gastric tube insertion | At 5 minutes
  Ease of passage of a gastric tube as: easy, difficult or impossible
Incidence of perioperative complications | 2 hours
  number of patients with adverse events: Airway obstruction, desaturation, Aspiration, oropharyngeal trauma, sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Lopez, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Ambulatory Surgery, Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain